CLINICAL TRIAL: NCT03308058
Title: Feasibility of a Touch Screen Computer Based Breast-feeding Educational Support Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0430-12-EP
Record Dates: First submitted 2012-10-30; First posted 2017-10-12 (Actual); Results first posted 2019-06-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Pregnancy Related
Keywords: Breastfeeding Rural Hispanic Pregnant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Breastfeeding Computer education (Experimental): Breastfeeding Computer education
  Interventions: Behavioral: Breastfeeding computer education
- Printed Educational material (No Intervention): Printed educational material

INTERVENTIONS:
Behavioral: Breastfeeding computer education — Breastfeeding computer education
  Arms: Breastfeeding Computer education

SUMMARY:
Breastfeeding has many positive and long lasting impacts on the health of infants and mothers. The investigators propose to develop a bilingual touch screen computer based breastfeeding educational support program to promote breastfeeding among Hispanic rural women living in Scottsbluff area of rural Nebraska. An interactive, tailored, touch screen, bilingual breastfeeding educational program will be developed to deliver breastfeeding education to enhance partial or exclusive breastfeeding. An experimental two-group repeated measures design will be utilized. Ninety four prenatal Hispanic rural women aged 15 years and above will be enrolled and randomly assigned to either the intervention (computer based program, N=47) or attention control (printed educational material, N=47) groups at the Regional West Medical Center in Scottsbluff. Information gathered will include socio-demographics, familiarity with use of technology and health literacy assessment. Process variables measured will include breast-feeding knowledge and breast-feeding self-efficacy. Primary and secondary outcomes include breast-feeding duration in binary categories (partial or exclusive) and number of sick baby medical visits and months of illnesses. All assessments will be done at baseline, days 3 and 7, weeks 2 and 6 and months 3 and 6 in both the intervention and attention intervention groups. The current proposed study may help advance our understanding to use health information technology as a medium to disseminate bilingual health education programs in rural settings. This exploratory study will lay a foundation for a larger multicenter randomized controlled clinical trial to evaluate the impact of computer based educational intervention to promote sustainability of breastfeeding among women across diverse settings.

DETAILED DESCRIPTION:
Two separate focus groups one in English and Spanish will be performed with six Hispanic rural women with history of previous pregnancy will be enrolled at the Regional West Medical Center (RWMC), Scottsbluff, NE. The focus group of 2 hours duration will be performed at the antenatal clinic at RWMC during months 2 and 3 of the study. The focus group will help examine factors that affect the decision to continue breast-feeding in pregnant Hispanic rural women and will guide development of bilingual (English and Spanish) breast-feeding educational modules during months 4 and 5 of the study. Dr. Aguirre and Ms. Salazar will be responsible for subject recruitment, focus group assessments and would act as a moderator and respond to questions and comments during the focus groups. The focus group interviews, analysis and development of breast-feeding educational modules in English and Spanish will be finalized during the first 5 months of the study. The focus group sessions will be audio recorded and stored in a locked cabinet. The sessions recordings will be destroyed at the end of the research study.

Computer-based Breast-Feeding Educational Support Program: The investigators will modify existing touch screen, computer based interactive Patient Education and Motivation Tool (PEMT) to deliver bilingual, breast-feeding educational support program. The existing PEMT platform allows users to dynamically change the educational content either to English or Spanish. The modification of the existing PEMT will occur during months 5-7 and will include several stages:

(i) PEMT modification design (ii) Tailoring (iii) Expert Pretesting using Heuristic evaluation (iv) Usability and User Testing

Intervention and Evaluation:

The subjects will be randomly enrolled using a 1:1 method with every other subject enrolled randomized to either the control or intervention group, at RWMC, Scottsbluff. Eligible individuals, who will meet the inclusion criteria, will be assigned into either intervention (bilingual Computer based Breast-feeding Educational Support program) or attention control (bilingual breast-feeding printed educational material) groups using a computer generated random id during the subject's prenatal visit (i.e. anytime during last six weeks of their pregnancy). Once randomized, baseline information will be gathered in both the groups.

The difference between the two study groups is that subjects in the intervention (bilingual Computer based Breast-feeding Educational Support program) will record their baseline assessment on a computer and receive tailored breast-feeding education compared to the attention control (bilingual printed breast-feeding educational materials) who will record their baseline information on paper and receive printed breast-feeding educational material. Using self-reported responses of the individuals in the intervention group (bilingual computer based breast-feeding educational support program), the decision logic and algorithm will process the information and deliver tailored breast-feeding educational messages in varied multimedia formats using a combination of text, images, and animations to account for the literacy levels of the subjects.

Appropriate feedback will be given in the form of reinforced educational messages and encouragement and motivational prompts for those using the computer based program. Educational session in both the groups will last for 30 minutes. The first educational session will be performed during the postpartum period, one day before the discharge from the hospital followed by week 6, months 3 and 6. Specific individualized interventions, especially during the initial critical 2-6 week period, are needed to prevent deterioration in intention levels for breast-feeding for 6 months and breast-feeding self-efficacy levels within the first 2 weeks postpartum which could lead to the decision to discontinue breast-feeding. Subjects in both the groups will be given telephone reminders for follow up educational sessions. The touch screen computer based Breast-feeding Educational Support program will be placed on a mobile cart in the outpatient clinic of the RWMC, Scottsbluff for the duration of the study and will be collected after the completion of the research.

There will be no repercussions to subjects since the touch screen computers will be placed at the RWMC and will be used by the subjects enrolled in the study at this site. A web based version will also be available for an ongoing support to subjects in the intervention group. A research assistant will be available to guide the subjects in both the intervention (during the use of the tablet pc program) and the control groups (printed educational material) if needed. The breast-feeding educational modules and data collection instruments will be both in English and Spanish.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic females age 15 years and above
* Pregnant
* Agreeing to participate in the study
* Understand spoken English
* Telephone at home
* Available for follow-up interview.

Exclusion Criteria:

* mental and physical challenge that makes it difficult to use the touch based computer program
* unavailability for telephone follow-up and
* involvement in other clinical trials or protocols related to breastfeeding.

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2012-10-18 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Wilhelm, PhD, Study Chair — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Regional West Medical Center, Scottsbluff, Nebraska, United States

REFERENCES:
- [Background] Thompson DA, Joshi A, Hernandez RG, Jennings JM, Arora M, Ellen JM. Interactive nutrition education via a touchscreen: is this technology well received by low-income Spanish-speaking parents? Technol Health Care. 2012;20(3):195-203. doi: 10.3233/THC-2012-0669. PMID 22735734
- [Background] Thompson DA, Joshi A, Hernandez RG, Bair-Merritt MH, Arora M, Luna R, Ellen JM. Nutrition education via a touchscreen: a randomized controlled trial in Latino immigrant parents of infants and toddlers. Acad Pediatr. 2012 Sep-Oct;12(5):412-9. doi: 10.1016/j.acap.2012.03.020. Epub 2012 Jun 7. PMID 22682718
- [Background] Joshi A, Weng W, Lichenstein R, Arora M, Sears A. Prospective tracking of a pediatric emergency department e-kiosk to deliver asthma education. Health Informatics J. 2009 Dec;15(4):282-95. doi: 10.1177/1460458209345899. PMID 20007653
- [Background] Joshi A, Arora M, Dai L, Price K, Vizer L, Sears A. Usability of a patient education and motivation tool using heuristic evaluation. J Med Internet Res. 2009 Nov 6;11(4):e47. doi: 10.2196/jmir.1244. PMID 19897458
- [Background] Joshi A, Lichenstein R, Rafei K, Bakar A, Arora M. A pilot study to evaluate self initiated computer patient education in children with acute asthma in pediatric emergency department. Technol Health Care. 2007;15(6):433-44. PMID 18057566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 46 mothers included in the study.
Groups:
- Computer Based Breast-feeding Education Group: This group of mothers received the book of breastfeeding modules and electronically the web based breast feeding educational support program
- Control Group: This group received the booklet format of the breast feeding educational support program
Period: Overall Study
Arm/Group | Computer Based Breast-feeding Education Group | Control Group
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Printed Educational Material: Printed educational material only
- Total: Total of all reporting groups
Arm/Group | Breastfeeding Computer Education | Printed Educational Material | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 23 | 46
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Breastfeeding Assessment
Description: Questionnaire Breastfeeding duration (Specify time) __________
Time Frame: 0-6 months
Population: no other primary or secondary measures to report
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Computer Based Breast-feeding Education Group | Control Group
Number analyzed (Participants) | 23 | 23
days | 121.2 (65.9) | 120.3 (61.8)

ADVERSE EVENTS:
Time Frame: 6 months per participant
Arm/Group | Computer Based Breast-feeding Education Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI, who is no longer with UNMC must approve all publications and make the sponsor AHRQ aware of them.

This is restrictive since he is now in New York and the study and data were and are in Nebraska.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT03308058/Prot_SAP_000.pdf